CLINICAL TRIAL: NCT03783494
Title: Target-controlled Infusion With Propofol in the Emergency Department : a Prospective Study on 45 Adult Patients
Acronym: SIVOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-PP-04
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Joint Dislocation; Limb Fracture
Keywords: ED; dislocation reduction; emergency department; TCI; Target-controlled infusion; sedation; fracture reduction
MeSH Terms: conditions — Joint Dislocations; Emergencies | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target-controlled infusion (TCI) (Experimental): Target-controlled infusion (TCI) with propofol up to 5.5µg/ml during an anticipated average maximal time of 15 minutes
  Interventions: Drug: Target control infusion with propofol

INTERVENTIONS:
Drug: Target control infusion with propofol — Target control infusion with propofol for patients with indications of sustaining very painful orthopedic emergency emergent procedures

SUMMARY:
Procedural sedation is an emergency medicine technique that provides a brief, deep sedation in order to perform very painful emergency emergent procedures such as displaced fracture or dislocated joints reduction. Propofol is recommended for this purpose, injected administered in slow IV bolus injections according to the technique known as manual titration. But despite this precaution, temporarily excessive sedation can happen, and a side effect can appear (arterial hypotension or respiratory depression). Target-controlled infusion (TCI) is an anesthesia technique that permits to obtain a precise constant and stable concentration of medication, boluses volumes of injection being calculated and delivered automatically by an electric syringe equipped with a software obedient to existing pharmacokinetic models. In the operating room, Ffor anesthetic induction, maintenance and awakening, respectively, in the operating room, the brain concentrations of propofol range respectively from 2 to 6 μg/mL, 2 to 4 μg/mL, and between 0.8 and 1.2 μg/mL, respectively. Since TCI has never been used in emergency departments (ED), the brain propofol concentrations which are necessary for sedation and awakening of the patient are not known and must be determined experimentally.

In this single-center, prospective, interventional study, safety and feasibility of TCI will be studied in one ED with the primary objective of determining the brain propofol concentrations necessary to reach the an optimal sedation in for patients with indications of sustaining very painful orthopedic emergency emergent procedures

DETAILED DESCRIPTION:
Procedural sedation is an emergency medicine technique that provides a brief, deep sedation in order to perform very painful emergency emergent procedures such as displaced fracture or dislocated joints reduction. For this purpose, propofol is a remarkable sedative agent for its very short elimination half-life, antiemetic property and myorelaxant effects. It is recommended to inject administer it in slow IV boluses injections according to the technique known as manual titration, but despite this precaution, temporarily excessive sedation can happen, and a side effect appear (arterial hypotension or respiratory depression).

Target-controlled infusion (TCI) is an anesthesia technique that permits to obtain a precise constant and stable concentration of medication, boluses volumes of injection being calculated and delivered automatically by an electric syringe equipped with a software obedient to existing pharmacokinetic models.

The age, size and weight of the patient are filledentered, then the syringe delivers the volume which is necessary and sufficient to reach and maintain the target concentration chosen by the practitioner. For anesthetic induction in the operating room, the brain concentrations of propofol used range from 2 to 6 μg/mL, then the general anesthesia maintenance is obtained with 2 to 4 μg/mL, and the patient awakening usually happens between 0.8 and 1.2 μg/mL. Since TCI has never been used in emergency departments (ED), the brain propofol concentrations which are necessary for sedation and awakening of the patient are not known and must be determined experimentally.

In this single-center, prospective, interventional study, safety and feasibility of TCI will be studied in an ED with the primary objective of determining the brain propofol concentrations necessary to reach the an optimal sedation in for patients with indications ofsustaining very painful orthopedic emergency emergent procedures. As secondary objectives, we will study the characteristics of sedations obtained (level, delays, lengths); the Delays, lengths and levels of sedation obtained, overall delivered doses of propofol administered; the , nature, appearance delays and lengths of potential adverse events (AE) related to procedural sedation, particularly complications related to procedural sedation, and necessary interventions necessary to handle these AE., will be studied as secondary objectives

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or more
* Affiliated or beneficiary of a French health insurance system
* Indication of procedural sedation, by the emergency department physician in the context of the management of for a patient with an orthopedic lesion requiring a potentially painful emergentcy therapeutic actionprocedure (reduction of a joint dislocation or realignment of a limb displaced fracture)
* For women :

  * at childbearing age : effective contraception (oral, intra-uterine device or condoms)
  * postmenopausal : amenorrhea for at least 12 month before the inclusion day
  * objective infertility (diagnosis or surgically)
* Signed free informed consent or inclusion in the context of an emergency situation

Exclusion Criteria:

* Patient of more than 18 under legal protection or deprivation of liberty measures
* Ongoing pregnancy or breastfeeding women
* Patient with the incapacity to give his free informed consent, excepted if the incapacity is induced by the context of the emergency situation (inclusion in the context of an emergency situation)
* Known hypersensitivity to propofol or one of the excipients, egg, sojasoya or peanuts
* ASA comorbidity score of 4 or more
* Heart, respiratory, renal or hepatic failure
* Epilepsy
* Lipid metabolism disorder
* Mitochondrial disease
* Hemodynamic instability, multiple traumatism
* Elevated intracranial tension
* Drug or alcohol intoxication
* Simultaneous participation to another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Propofol brain concentration | Between the beginning of sedation (T0) and the beginning of the orthopedic procedure (T_Ramsay5)
  Propofol brain concentration necessary for the patient to reach a Ramsay score of 5 (optimal sedation) (Ce_Ramsay5)

SECONDARY OUTCOMES:
Delay between the beginning of sedation (T0) and the beginning of the orthopedic procedure (T_Ramsay5) | the delay is the outcome, T_Ramsay5 (up to an anticipated average maximal time of 15 minutes after T0)]
  the delay is the outcome, T_Ramsay5 (up to an anticipated average maximal time of 15 minutes after T0)]
Propofol brain concentration when the patient spontaneously reopen his eyes (Ce_OuvertureYeux) | Time after T0 when the patient spontaneously reopen his eyes (up to an anticipated average maximal time of 30 minutes after T0)
  Propofol brain concentration when the patient spontaneously reopen his eyes after the orthopedic procedure has been realized, the TCI syringe been switched off, and the immobilization been placed (Ce_OuvertureYeux)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien LEMOEL, PhD, Principal Investigator — Emergency Department, Universitary Hospital of Nice
Locations (1):
- Emergency Department, Nice, France

IPD SHARING:
Plan to Share IPD: No